CLINICAL TRIAL: NCT03261700
Title: Recovering From Intimate Partner Violence Through Strengths and Empowerment (RISE): Tailoring and Evaluating a Patient-Centered Counseling Intervention for Women Veterans
Brief Title: Recovering From Intimate Partner Violence Through Strengths and Empowerment (RISE)
Acronym: RISE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: VA Boston Healthcare System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIR 16-062; 1I01HX002178-01A1 (NIH)
Record Dates: First submitted 2017-08-17; First posted 2017-08-25 (Actual); Results first posted 2023-03-30 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Intimate Partner Violence; Self-efficacy
Keywords: women Veterans; interpersonal violence

STUDY DESIGN:
Intervention Model Description: For the RCT (Aim 3), participants will be randomized to RISE or an information and referral condition.
Masking Description: Open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- RISE (Experimental): This provider- administered brief- counseling intervention program will increase Women Veteran?s self- efficacy in addressing violence in their current or past relationships. The variable length (up to six- session) modular-based intervention aims at providing resources for WVs in the relevant domains of: 1) safety planning, 2) education on health effects of IPV, 3) improving coping and self- care and red flags, 4) enhancing social support, 5) making difficult decisions, and 5) connecting with resources.
  Interventions: Behavioral: RISE
- Information and referral condition (Active Comparator): This brochure-based intervention includes education about IPV, health effects of IPV, resources and referral options to address a wide-array of health and social issues associated with IPV, and safety planning. Participants randomized to this arm are offered resources and referrals to VA and community resources.
  Interventions: Other: Information and referral condition

INTERVENTIONS:
Behavioral: RISE — This provider- administered brief- counseling intervention program will increase Women Veteran's self- efficacy in addressing violence in their current or past relationships. The variable length (up to six- session) modular-based intervention aims at providing resources for WVs in the relevant domains of: 1) safety planning, 2) education on health effects of IPV and red flags, 3) improving coping and self- care, 4) enhancing social support, 5) making difficult decisions, and 5) connecting with resources.
  Other Names: Recovering from IPV through Strengths and Empowerment
  Arms: RISE
Other: Information and referral condition — Participants randomized to this arm will receive a brochure-based intervention, consisting of education, support and problem solving, safety planning as well as resources and referrals to address an array of health and social issues associated with IPV (including in VA and the community).
  Other Names: Control condition
  Arms: Information and referral condition

SUMMARY:
Intimate partner violence (IPV) is a major health concern for women Veterans. IPV is associated with numerous physical and mental health conditions. VHA is implementing IPV screening programs to identify female patients who experience past-year IPV. Despite strong evidence that screening increases detection of IPV, less is established about how to intervene following IPV disclosure in health care settings, in order to improve health outcomes. Existing healthcare-based interventions result in minimal effects on health and well-being, likely because they are too brief and generic.

In response, the PI has developed Recovering from IPV through Strengths and Empowerment (RISE), based on the IPV-related health care needs and preferences of women Veterans. RISE is designed to be delivered in primary care and is an individualized, variable-length, modular-based intervention that addresses

* safety planning;
* education on the health effects of IPV and warning signs;
* increasing coping skills and self-care;
* enhancing social support;
* making difficult decisions; and
* connecting with resources. This study is aimed at refining and evaluating RISE for use with female VA patients who have experienced past-year IPV. This brief counseling intervention is intended to be administered in conjunction with primary care, as this is a frequent point of healthcare contact for women Veterans and where disclosure of IPV is most prevalent.

DETAILED DESCRIPTION:
Women are the fastest growing group of VHA patients, with their population recently increasing by 80%. Women Veterans (WV's) are at higher risk for IPV than their non-Veteran peers, with that 1 in 3 WVs report lifetime IPV, compared to 1 in 4 women in the general U.S. population. Research reports up to 30% of WVs experience past-year IPV. As a result, WVs are considered an important population for IPV screening and counseling interventions. In response, VHA Women's Health Services (WHS) and the IPV Assistance Program of Care Management and Social Work Services (CMSWS) are implementing IPV screening programs for women and are seeking an effective intervention to implement into care. Extant brief counseling interventions for IPV result in minimal effects on patients' health and safety. A recent review of IPV screening trials highlighted insufficient intensity of post-disclosure counseling interventions, concluding that existing interventions are too brief, unstructured, and generic. Such minimal intervention effects of the current standard of care have led leaders in the field to call for the development and testing of new and more comprehensive IPV interventions, especially for delivery in conjunction with primary care. The Recovering from IPV through Strengths and Empowerment (RISE) intervention fills this need.

The PI, a clinical psychologist and health services researcher with expertise in and national recognition for IPV research and care, has developed an innovative IPV intervention to respond to this need. Recovering from IPV through Strengths and Empowerment (RISE) is based on the healthcare needs and preferences of WVs who have experienced IPV. RISE was developed using rigorous methods, building on the evidence base from the applicant's HSR&D CDA and on input of VHA primary care and behavioral health experts. RISE is based on empowerment, a highly relevant intervention model for women who experience IPV. It is an individualized, variable-length, modular-based intervention addressing key factors:

* safety planning,
* educating about the health effects of IPV and warning signs,
* improving coping and self-care,
* enhancing social support,
* making difficult decisions, and
* connecting with resources. RISE is rooted in empowerment and incorporates aspects of Motivational Interviewing, an evidence-based approach designed to facilitate behavior change that is widely used in VHA for numerous health issues.

This timely research project addresses the critical gap in current IPV care. It will refine and formally evaluate RISE using established methods for rapid and efficient effectiveness testing, including a Hybrid 1 randomized clinical trial (RCT) to evaluate RISE that simultaneously gathers information on barriers to and facilitators of implementation. The study is guided by the first two phases of the Replicating Effective Programs (REP) framework, pre-conditions and pre-implementation. These phases emphasize tailoring interventions with stakeholder input and iterative cycles of pilot testing within routine practice conditions. Use of the REP framework will maximize the likelihood that RISE-should its effectiveness be demonstrated-can easily be integrated into routine care in VHA.

The Specific Aims of this study are as follows:

1. Tailor and refine RISE to accommodate differences in service structures and personnel in different primary care settings through input from a Stakeholder Advisory Board, focus groups with WVs (four groups; n=24-32), and qualitative interviews with providers (n=24).
2. Conduct a formative evaluation of RISE with WVs (n=up to 20) to inform the development of a user-friendly, tailored implementation protocol and intervention manual.
3. Examine the effects of RISE on WVs' (n=60) individual psychosocial outcomes (e.g., empowerment, self-efficacy, health symptoms, service use, and quality of life) in an RCT that compares RISE to an information/referral condition.

3a. Evaluate the feasibility and acceptability of RISE in the context of the RCT.

This study provides the groundwork to examine the effectiveness of RISE. The data will be used to demonstrate whether the effects of RISE appear promising to support a future-large scale effectiveness-implementation RCT, including the range of effect sizes that would be reasonable to expect in a future trial.

The project was originally conducted at two Women's Health Practice-Based Research Network (PBRN) sites that have adopted IPV screening - the Women's Health Centers (WHC) at VA Boston Healthcare System and VA Connecticut Healthcare System. RCT study enrollment was discontinued at VA Connecticut in July 2019 due to low enrollment. The VA Boston Healthcare System serves as the sole site for data collection from July 2019 on and is the sourced of the RCT data.

The COVID-19 pandemic resulted in modifications to IRB protocol to switch from in-person enrollment, assessments and sessions. There were several women actively involved in the trial during the initial shut-down. New recruitment and enrollment were temporarily hauled during early months of COVID-19, with virtual enrollment beginning as of July 2020.

Recruitment and enrollment were completed in September 2020 because the enrollment goals were met and the planned sample size was obtained (N=60).

ELIGIBILITY:
Inclusion Criteria:

Participants will be eligible to participate if they:

* Self-identify as a woman
* Are at least 18 years of age
* A patient at VA Boston Healthcare System
* Self- reported that they have experienced past-year physical, sexual, or psychological IPV
* Ability to understand study procedures in English
* Not exhibiting symptoms of mania or psychosis
* Not actively in suicidal crisis warranting imminent hospitalization

Exclusion Criteria:

* Any violation of inclusion criteria

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Self-identify as female
Enrollment: 60 (Actual)
Dates: Start 2018-10-22 (Actual); Primary Completion 2020-11-23 (Actual); Study Completion 2020-11-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine M. Iverson, PhD MA BA, Principal Investigator — VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA
Locations (1):
- VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dardis CM, Dichter ME, Iverson KM. Empowerment, PTSD and revictimization among women who have experienced intimate partner violence. Psychiatry Res. 2018 Aug;266:103-110. doi: 10.1016/j.psychres.2018.05.034. Epub 2018 May 30. PMID 29859496
- [Background] Grillo AR, Danitz SB, Dichter ME, Driscoll MA, Gerber MR, Hamilton AB, Wiltsey-Stirman S, Iverson KM. Strides Toward Recovery From Intimate Partner Violence: Elucidating Patient-Centered Outcomes to Optimize a Brief Counseling Intervention for Women. J Interpers Violence. 2021 Aug;36(15-16):NP8431-NP8453. doi: 10.1177/0886260519840408. Epub 2019 Apr 17. PMID 30994401
- [Background] Iverson KM, Dardis CM, Grillo AR, Galovski TE, Pogoda TK. Associations between traumatic brain injury from intimate partner violence and future psychosocial health risks in women. Compr Psychiatry. 2019 Jul;92:13-21. doi: 10.1016/j.comppsych.2019.05.001. Epub 2019 May 14. PMID 31203176
- [Background] Danitz SB, Stirman SW, Grillo AR, Dichter ME, Driscoll M, Gerber MR, Gregor K, Hamilton AB, Iverson KM. When user-centered design meets implementation science: integrating provider perspectives in the development of an intimate partner violence intervention for women treated in the United States' largest integrated healthcare system. BMC Womens Health. 2019 Nov 27;19(1):145. doi: 10.1186/s12905-019-0837-8. PMID 31771557
- [Background] Iverson KM, Danitz SB, Driscoll M, Vogt D, Hamilton AB, Gerber MR, Wiltsey Stirman S, Shayani DR, Suvak MK, Dichter ME. Recovering from intimate partner violence through Strengths and Empowerment (RISE): Development, pilot testing, and refinement of a patient-centered brief counseling intervention for women. Psychol Serv. 2022;19(Suppl 2):102-112. doi: 10.1037/ser0000544. Epub 2021 Jun 10. PMID 34110870
- [Result] Iverson KM, Danitz SB, Shayani DR, Vogt D, Stirman SW, Hamilton AB, Mahoney CT, Gerber MR, Dichter ME. Recovering From Intimate Partner Violence Through Strengths and Empowerment: Findings From a Randomized Clinical Trial. J Clin Psychiatry. 2021 Nov 23;83(1):21m14041. doi: 10.4088/JCP.21m14041. PMID 34813687
- [Result] Shayani DR, Danitz SB, Low SK, Hamilton AB, Iverson KM. Women Tell All: A Comparative Thematic Analysis of Women's Perspectives on Two Brief Counseling Interventions for Intimate Partner Violence. Int J Environ Res Public Health. 2022 Feb 22;19(5):2513. doi: 10.3390/ijerph19052513. PMID 35270204
- [Result] Davin KR, Dardis CM, Barth MR, Iverson KM. Prospective mental health effects of intimate partner stalking among women veterans. Psychol Trauma. 2022 Jul;14(5):751-758. doi: 10.1037/tra0001144. Epub 2021 Nov 4. PMID 34735188
- [Result] Iverson KM, Dardis CM, Cowlishaw S, Webermann AR, Shayani DR, Dichter ME, Mitchell KS, Mattocks KM, Gerber MR, Portnoy GR. Effects of Intimate Partner Violence During COVID-19 and Pandemic-Related Stress on the Mental and Physical Health of Women Veterans. J Gen Intern Med. 2022 Sep;37(Suppl 3):724-733. doi: 10.1007/s11606-022-07589-z. Epub 2022 Aug 30. PMID 36042090
- [Result] Webermann AR, Dardis CM, Iverson KM. The role of general self-efficacy in intimate partner violence and symptoms of posttraumatic stress disorder among women veterans. J Trauma Stress. 2022 Jun;35(3):868-878. doi: 10.1002/jts.22794. Epub 2022 Jan 31. PMID 35099821

RESULTS

PARTICIPANT FLOW:
Groups:
- RISE: This provider- administered brief- counseling intervention program will increase Women Veterans self- efficacy and personal empowerment in addressing violence in their current or past relationships. The variable length (up to six- session) modular-based intervention aims at providing resources for women veterans in the relevant domains of: 1) safety planning, 2) education on health effects of IPV, 3) improving coping and self- care and red flags, 4) enhancing social support, 5) making difficult decisions, and 5) connecting with resources and moving forward.
  RISE: This provider- administered brief- counseling intervention program will increase Women Veteran's self- efficacy in addressing violence in their current or past relationships. The variable length (up to six- session) modular-based intervention aims at providing resources for WVs in the relevant domains of: 1) safety planning, 2) education on health effects of IPV and red flags, 3) improving coping and self- care, 4) enhancing social support, 5) making difficult decisions, and 5) connecting with resources.
- Enhanced Care as Usual Condition: This brochure-based intervention includes education about IPV, health effects of IPV, resources and referral options to address a wide-array of health and social issues associated with IPV, and safety planning. Participants randomized to this arm are offered resources and referrals to VA and community resources.
  Information and referral condition: Participants randomized to this arm will receive a brochure-based intervention, consisting of education, support and problem solving, safety planning as well as resources and referrals to address an array of health and social issues associated with IPV (including in VA and the community).
Period: Overall Study
Arm/Group | RISE | Enhanced Care as Usual Condition
Started | 30 | 30
Completed | 29 (1 participant did not attend either the 10 or 14 week follow-up assessment and thus is not included in primary intent-to-treat (ITT) analyses. The participant was not able to participate due to COVID-19 related stressors.) | 30
Not Completed | 1 | 0
Not completed — The participant was not able to participate due to COVID-19 related stressors. | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RISE | Enhanced Care as Usual Condition | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.7 (10.8) | 40.5 (13.0) | 39.1 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 30 | 60
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 5 | 12
  Not Hispanic or Latino | 23 | 25 | 48
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 8 | 5 | 13
  White | 17 | 16 | 33
  More than one race | 3 | 5 | 8
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30 | 30 | 60
Sexual orientation [Count of Participants; unit: Participants]
  Heterosexual | 19 | 24 | 43
  Lesbian/Gay | 3 | 1 | 4
  Bisexual | 5 | 4 | 9
  Pansexual | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Empowerment Via the Personal Progress Scale Revised
Description: Measures change in sense of personal empowerment; minimum value = 28 and maximum score = 196; higher scores indicate higher personal empowerment
Time Frame: Baseline,10-week follow-up, and 14-week follow-up assessments
Population: Intent-to-treat (ITT) sample
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | RISE | Enhanced Care as Usual Condition
Number analyzed (Participants) | 29 | 30
score on a scale
  Baseline | 129.82 [121.91 to 137.73] | 132.25 [123.64 to 140.87]
  10-Week Follow-up | 146.13 [137.80 to 154.46] | 137.24 [129.85 to 144.63]
  14-Week Follow-up | 148.07 [139.62 to 156.52] | 137.66 [130.15 to 145.17]
Statistical Analysis 1: Comparison: RISE vs Enhanced Care as Usual Condition; Comparison of groups on Empowerment via the Personal Progress Scale Revised; Test type: Superiority; p < .05, Mixed Models Analysis

2. Primary Outcome: Self-efficacy Via the General Self-Efficacy Scale
Description: This scale is a self-report of change in general self-efficacy; minimum score = 4 and maximum score = 40; higher scores indicate higher self-efficacy
Time Frame: Baseline, 10-week follow-up, and 14-week follow-up assessments
Population: Intent-to-Treat (ITT) sample
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | RISE | Enhanced Care as Usual Condition
Number analyzed (Participants) | 29 | 30
score on a scale
  Baseline | 28.7 [27.04 to 30.36] | 29.90 [27.98 to 31.82]
  10-Week Follow-up | 33.33 [31.75 to 34.91] | 30.66 [29.01 to 32.31]
  14-Week Follow-up | 34.07 [32.53 to 35.61] | 30.52 [28.95 to 32.09]
Statistical Analysis 1: Comparison: RISE vs Enhanced Care as Usual Condition; Comparison of groups on self-efficacy via the General Self-Efficacy Scale; Test type: Superiority; p < .05, Mixed Models Analysis

3. Primary Outcome: Valued Living Questionnaire
Description: Measures change in valued living, and congruence between stated values and past-week valued behavior; Composite scores range from 10 (minimum) to 100 (maximum). Higher scores reflect higher valued living (i.e., an indicator of higher quality of life)
Time Frame: Baseline, 10-week follow-up, and 14-week follow-up assessments
Population: Intent-to-Treat (ITT) sample
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | RISE | Enhanced Care as Usual Condition
Number analyzed (Participants) | 29 | 30
score on a scale
  Baseline | 49.88 [42.97 to 56.79] | 48.88 [42.87 to 54.89]
  10-Week Follow-up | 63.27 [56.68 to 69.86] | 53.44 [46.86 to 60.02]
  14-Week Follow-Up | 60.96 [52.62 to 69.30] | 57.23 [50.51 to 63.95]

4. Primary Outcome: Patient Activation Measure (PAM-13)
Description: Measures change in patient engagement in needed health care; scores are transferred to a theoretical 0-100 scale; higher scores indicate higher patient activation.
Time Frame: Baseline, 10-week follow-up, and 14-week follow-up assessments
Population: Intent-to-Treat (ITT) Sample
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | RISE | Enhanced Care as Usual Condition
Number analyzed (Participants) | 29 | 30
score on a scale
  Baseline | 65.89 [59.19 to 72.58] | 64.62 [58.64 to 70.61]
  10-week follow-up assessment | 76.5 [69.49 to 83.51] | 69.24 [64.30 to 74.19]
  14-week follow-up assessment | 75.5 [67.87 to 83.13] | 70.12 [65.50 to 74.65]

5. Secondary Outcome: PTSD Checklist for DSM-5
Description: Measures change in DSM-5 PTSD symptom severity. Scores range from 0-80; higher scores reflect higher/worse PTSD symptoms.
Time Frame: Baseline, 10-week follow-up, and 14-week follow-up assessments
Population: Intent-to-Treat (ITT) Sample
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | RISE | Information and Referral Condition
Number analyzed (Participants) | 29 | 30
score on a scale
  Baseline | 41.92 [35.98 to 47.85] | 39.97 [34.20 to 45.73]
  10-week assessment | 29.97 [22.69 to 36.72] | 36.97 [31.25 to 42.68]
  14-week assessment | 32.73 [25.11 to 40.35] | 32.13 [25.61 to 38.65]

6. Secondary Outcome: Center for Epidemiological Studies-Depression Scale
Description: Measures change in depressive symptoms; This measure ranges from 0-60; higher scores reflect (worse) higher levels of symptoms
Time Frame: Baseline, 10-week follow-up, and 14-week follow-up assessments
Population: Intent-to-treat (ITT) sample
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | RISE | Enhanced Care as Usual Condition
Number analyzed (Participants) | 29 | 30
score on a scale
  Baseline | 27.21 [23.38 to 31.04] | 24.50 [20.29 to 28.71]
  10-week follow-up | 19.59 [14.84 to 24.34] | 22.76 [19.36 to 26.16]
  14-week follow-up | 21.12 [15.77 to 26.47] | 19.72 [15.32 to 24.12]

7. Secondary Outcome: SF-12 Health Survey
Description: Measures change in physical-health related quality of life. Specifically, quantitative ratings of overall physical health functioning were rated on a Likert scale of 1-5 (1 = excellent, 2 = very good, 3 = good, 4 = fair, 5 = poor).
Time Frame: Baseline, 10-Week follow-up, and 14-Week follow-up Assessments
Population: Intent-to-treat (ITT) sample
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | RISE | Enhanced Care as Usual Condition
Number analyzed (Participants) | 29 | 30
score on a scale
  Baseline | 3 (.87) | 3 (.77)
  10-Week Follow-Up | 3 (.87) | 2 (.74)
  14-Week Follow-Up | 3 (.76) | 3 (.87)

8. Secondary Outcome: Conflict Tactic Scales Revised
Description: Measures change in overall number of different IPV acts over time (i.e., total count score). This measure ranges from 0-33; higher scores reflect higher levels of IPV (i.e., a worse outcome).
Time Frame: Baseline, 10-week follow-up, and 14-week follow-up assessments
Population: ITT sample
Measure: Mean (95% Confidence Interval); unit: units on a scale (count scores)
Arm/Group | RISE | Enhanced Care as Usual Condition
Number analyzed (Participants) | 29 | 30
units on a scale (count scores)
  Baseline | 11.17 [8.15 to 14.2] | 11.67 [9.14 to 14.2]
  10-Week Follow-up | 3.37 [2.20 to 4.54] | 4.93 [2.56 to 7.3]
  14-Week Follow-up | 3.34 [1.17 to 5.51] | 2.8 [1.76 to 3.84]

9. Secondary Outcome: Physical, Mental and Social Service Care Use
Description: Measures overall number of VA and non-VA health care visits (inclusive of physical, mental health, and social service use visits).
Time Frame: Baseline, 10-week follow-up, and 14-week follow-up assessments
Population: Intent-to-treat (ITT) sample
Measure: Mean (95% Confidence Interval); unit: visits
Arm/Group | RISE | Enhanced Care as Usual Condition
Number analyzed (Participants) | 29 | 30
visits
  Baseline | 8.27 [6.31 to 10.23] | 7.03 [5.29 to 8.77]
  10-Week Follow-Up | 6.15 [4.44 to 7.86] | 6.24 [4.69 to 7.79]
  14-Week Follow-Up | 4.62 [3.18 to 6.05] | 4.93 [3.35 to 6.52]

10. Secondary Outcome: Client Services Questionnaire (CSQ-8)
Description: Measures satisfaction with treatment; Scores range from 8 to 32; higher scores reflect higher satisfaction with treatment (i.e., a better outcome)
Time Frame: 10-week follow-up assessment
Population: Intent-to-Treat (ITT) Sample
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RISE | Enhanced Care as Usual Condition
Number analyzed (Participants) | 29 | 30
score on a scale | 29.30 (2.78) | 25.07 (4.85)

11. Secondary Outcome: Patient Health Questionnaire
Description: Measures change in somatic and physical health symptoms; score ranges from 0 to 30, with higher scores representing higher levels of physical health problems
Time Frame: Baseline, 10-week follow-up, and 14-week follow-up assessments
Population: Intent-to-treat (ITT) sample
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | RISE | Enhanced Care as Usual Condition
Number analyzed (Participants) | 29 | 30
score on a scale
  Baseline | 12.52 [10.41 to 14.63] | 10.60 [9.03 to 12.16]
  10-Week Follow-Up | 11.37 [9.33 to 13.41] | 12.01 [10.27 to 13.75]
  14-Week Follow-Up | 11.42 [8.99 to 13.85] | 9.69 [8.01 to 11.36]

12. Secondary Outcome: Safety Behaviors Checklist
Description: Measures the present use of safety behaviors participants are currently using to protect themselves. Each of the 15 items of this measure corresponds to a specific safety behavior. Participant indicates whether they have used each behavior using a dichotomous response option (yes = 1; no = 0). Scores are summed, with total scores ranging from 0-15. Higher scores indicate a higher number of safety behaviors enacted.
Time Frame: Baseline, 10-week follow-up, and 14-week follow-up assessments
Population: Intent-to-treat (ITT) sample
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | RISE | Enhanced Care as Usual Condition
Number analyzed (Participants) | 29 | 30
score on a scale
  Baseline | 12.87 [11.97 to 13.77] | 12.94 [12.09 to 13.79]
  10-Week Follow-Up | 13.04 [11.59 to 14.49] | 12.39 [10.79 to 13.99]
  14-Week Follow-Up | 9.4 [6.85 to 11.95] | 12.34 [10.75 to 13.93]

13. Secondary Outcome: Connor-Davidson Resilience Scale
Description: Measures patient resilience; Scores range from 0-100,with higher scores reflecting higher resilience
Time Frame: Baseline, 10-week follow-up, and 14-week follow-up assessments
Population: Intent-to-treat (ITT) sample
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | RISE | Enhanced Care as Usual Condition
Number analyzed (Participants) | 29 | 30
score on a scale
  Baseline | 25.43 [23.28 to 27.59] | 24.1 [21.87 to 26.33]
  10-Week Follow-Up | 29.67 [27.24 to 32.09] | 26 [23.9 to 28.1]
  14-Week Follow-Up | 29.65 [26.9 to 32.41] | 26.07 [23.8 to 28.34]

14. Secondary Outcome: Depression Anxiety Stress Scale- Anxiety Subscale
Description: Measures anxiety symptom severity; Scores range from 0-42, with higher scores indicating higher levels of anxiety.
Time Frame: Baseline, 10-week follow-up, and 14-week follow-up assessments
Population: Intent-to-treat (ITT) sample
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | RISE | Enhanced Care as Usual Condition
Number analyzed (Participants) | 29 | 30
score on a scale
  Baseline | 25.11 [21.83 to 28.38] | 23.4 [20.68 to 26.12]
  10-Week Follow-Up | 22.67 [18.92 to 26.41] | 22.98 [20.72 to 25.24]
  14-Week Follow-Up | 23.58 [19.88 to 27.28] | 21.22 [19.02 to 23.42]

15. Secondary Outcome: Coping Strategies Inventory - Short Form
Description: Measures engagement coping skills; Scores range from 8-40, with higher score reflecting better coping
Time Frame: Baseline, 10-week follow-up, and 14-week follow-up assessments
Population: Intent-to-treat (ITT) sample
Measure: Mean (95% Confidence Interval); unit: mean score on a scale
Arm/Group | RISE | Enhanced Care as Usual Condition
Number analyzed (Participants) | 29 | 30
mean score on a scale
  Baseline | 26.42 [25.22 to 27.61] | 25.69 [24.66 to 26.71]
  10-Week Follow-Up | 27.30 [25.99 to 28.61] | 25.74 [24.71 to 26.78]
  14-Week Follow-Up | 26.92 [25.72 to 28.13] | 25.4 [24.5 to 26.30]

16. Secondary Outcome: Brief Semi-structured Interview to Assess Acceptability and Feasibility of the Intervention, With Perceived Helpfulness Rating.
Description: Semi-structured qualitative interview questions developed for the purpose of this study to assess participants' perceptions of the acceptability, with a particular item to assess overall helpfulness of the intervention. Specifically, quantitative ratings of overall helpfulness were rated on a Likert scale of 1-5 (1=highly helpful, 2 = somewhat helpful, 3 = neither helpful nor unhelpful, 4 = somewhat unhelpful, 5=highly unhelpful).
Time Frame: Assessed at 10-week follow-up or 14-week follow-up, values at the end of 14 weeks reported
Population: Intent-to-Treat sample with completed helpfulness ratings at the 10- or 14-week follow-up assessments. From the RISE condition, 26 participants completed this assessment at the 10-week follow-up, and the remaining 3 completed it at the 14-week follow-up. From the Information and Referral condition, 29 participants completed this assessment at the 10-week follow-up and 1 participant completed it at the 14-week follow-up. Thus, the data represents summed count scores for each endorsed answer.
Measure: Count of Participants; unit: Participants
Groups:
- RISE: This provider- administered brief- counseling intervention program will increase Women Veteran's self- efficacy in addressing violence in their current or past relationships. The variable length (up to six- session) modular-based intervention aims at providing resources for WVs in the relevant domains of: 1) safety planning, 2) education on health effects of IPV, 3) improving coping and self- care and red flags, 4) enhancing social support, 5) making difficult decisions, and 5) connecting with resources.
  RISE: This provider- administered brief- counseling intervention program will increase Women Veteran's self- efficacy in addressing violence in their current or past relationships. The variable length (up to six- session) modular-based intervention aims at providing resources for WVs in the relevant domains of: 1) safety planning, 2) education on health effects of IPV and red flags, 3) improving coping and self- care, 4) enhancing social support, 5) making difficult decisions, and 5) connecting with resources.
Arm/Group | RISE | Information and Referral Condition
Number analyzed (Participants) | 29 | 30
Participants
  'Highly helpful' | 23 | 16
  'Somewhat helpful' | 6 | 14
  'Neither helpful or unhelpful' | 0 | 0
  'Somewhat unhelpful' | 0 | 0
  'Highly unhelpful' | 0 | 0

ADVERSE EVENTS:
Time Frame: 10-14 weeks following enrollment
Arm/Group | RISE | Enhanced Care as Usual Condition
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 4/30 | 1/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RISE (N=30) | Enhanced Care as Usual Condition (N=30)
hospitalized for medical condition (General disorders) | 4 | 1 — Participants reported at the follow up assessment having been hospitalized for general medical conditions. These events were deemed by the IRB as not unexpected, not related to research participation, and involved no increased risk

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-05-12): https://cdn.clinicaltrials.gov/large-docs/00/NCT03261700/Prot_SAP_000.pdf
  • Informed Consent Form (2020-06-08): https://cdn.clinicaltrials.gov/large-docs/00/NCT03261700/ICF_001.pdf